CLINICAL TRIAL: NCT05206357
Title: A Single Arm, Open-Label, Phase 1b Trial of Epcoritamab in Pediatric Patients With Relapsed/Refractory Aggressive Mature B-cell Neoplasms
Brief Title: Study of the Adverse Events and Change in Disease State of Pediatric Participants (and Young Adults Between the Ages of 18-25) With Relapsed/Refractory Aggressive Mature B-cell Neoplasms Receiving Subcutaneous (SC) Injections of Epcoritamab
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20-429; 2021-004555-16 (EudraCT Number)
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Non-hodgkin Lymphoma
Keywords: Non-hodgkin Lymphoma; ABBV-GMAB-3013; Epcoritamab; Burkitt's or Burkitt-like Lymphoma/Leukemia; Diffuse Large B-cell Lymphoma; Aggressive Mature (CD20+) B-cell Lymphoma; Cancer; Relapsed/Refractory Aggressive Mature B-cell Neoplasms; EPCORE
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epcoritamab (Experimental): Participants will receive subcutaneous (SC) epcoritamab in 28 day cycles.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection (SC)
  Other Names: ABBV-GMAB-3013

SUMMARY:
The most common types of mature B-cell lymphomas (MBLs) in children are Burkitt lymphoma (BL) and diffuse large B-cell lymphoma (DLBCL). Initial treatment cures 90% - 95% of children with these malignancies, leaving a very small population of relapsed/refractory disease with a poor prognosis. The purpose of this study is to assess the safety and tolerability of epcoritamab in pediatric participants with relapsed/refractory aggressive mature B-cell neoplasms and young adult participants with Burkitt's or Burkitt-like lymphoma/leukemia. Adverse events and change in disease activity will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of relapsed/refractory aggressive mature B-cell neoplasms. Participants will receive subcutaneous (SC) of epcoritamab. Approximately 15 pediatric participants with a diagnosis of relapsed/refractory aggressive mature B-cell neoplasms and and young adult participants, ages of 18-25, with a diagnosis of Burkitt's or Burkitt-like lymphoma/leukemia will be enrolled at 50 sites globally.

Participants will receive subcutaneous epcoritamab in 28-day cycles. Participants will be followed for a minimum of 3 years after enrollment.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants >= 1 and < 18 years old at time of primary diagnosis with Burkitt's or Burkitt-like lymphoma/leukemia, diffuse large B-cell lymphoma (DLBCL), or other aggressive mature (CD20+) B-cell lymphomas. Participants up to 25 years of age with Burkitt's or Burkitt-like lymphoma/leukemia are also eligible.
* Disease pathologically confirmed (tumor tissue) by local testing.
* Relapsed or primary refractory disease meeting any of the following criteria:

  * Progressive disease at any time during second-line chemoimmunotherapy (CIT).
  * Best response of stable disease (SD) after a minimum of 2 cycles of second-line CIT.
  * Best response of partial response (PR) after a minimum of 3 cycles of second-line CIT.
  * Complete Response (CR) after a minimum of 3 cycles of second-line CIT therapy but unfit or ineligible for consolidation with cell therapy.
  * Not in CR and unable to initiate or tolerate (i.e., must discontinue) second-line CIT.
  * Have received cell therapy (allogeneic or autologous transplant or chimeric antigen receptor T-cell (CAR-T) therapy) as consolidation but have not obtained or maintained a CR.
* Recovery from toxic effects of prior chemoimmunotherapy.
* Performance status by Lansky (< 16 years old at evaluation) or Karnofsky (>= 16 years old at evaluation) score >= 50 or Eastern Cooperative Oncology Group (ECOG) score <= 2 .
* Adequate bone marrow, hepatic, and renal function.

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma at screening as confirmed by screening magnetic resonance imaging (MRI)/computed tomography (CT)/positron emission tomography (PET) brain scans (participants with evidence of CNS disease only in the cerebrospinal fluid (CSF) will be eligible).
* Other malignancy requiring therapy.
* Currently receiving anti-cancer therapy, including chemotherapy (excluding intrathecal therapy), radiotherapy, small molecules, monoclonal antibodies, cell therapy, or other investigational agents.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 3 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Concentration (Cmax) | Up to Approximately Week 37
  Maximum observed concentration.
Area Under the Concentration Versus Time Curve (AUC) from Time 0 to Time of Last Measurable Concentration within the Dosing Interval (AUCtau) | Up to Approximately Week 37
  AUC from time 0 to time of last measurable concentration within the dosing interval.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Complete Response (CR) | Up to Approximately 1 Year
  CR is defined per the International Pediatric Non-Hodgkin Lymphoma Response Criteria as computed tomography (CT) or magnetic resonance imaging (MRI) reveals no residual disease or new lesions; Resected residual mass that is pathologically (morphologically) negative for disease (detection of disease with more sensitive techniques); bone marrow (BM) and cerebrospinal fluid (CSF) morphologically free of disease (detection of disease with more sensitive techniques).
Number of Participants with Event-free survival (EFS) | Up to Approximately 3 Years
  EFS will be defined as the number of days from screening to the date of disease progression, treatment failure, or death from any cause.
Number of Participants who Achieve Overall Survival (OS) | Up to Approximately 3 Years
  OS will be defined as the number of days from screening to the date of death from any cause.
Rate of Initiation of Stem Cell Transplantation or Chimeric Antigen Receptor T-cell (CAR-T) Therapy | Up to Approximately 1 Year
  Rate of initiation of stem cell transplantation or CAR-T therapy.
Percentage of Participants Achieving Overall Response (OR) | Up to Approximately 1 Year
  OR is assessed as the percentage of participants with an overall response.
Duration of response (DOR) | Up to Approximately 1 Year
  DOR is defined as the time between the date of first response to the date of the first documented tumor progression or death due to any cause, whichever comes first.
Duration of CR (DOCR) | Up to Approximately 1 Year
  DOCR is defined as the time between the date of first CR to the date of the first documented tumor progression or death due to any cause, whichever comes first.
Percentage of Participants Achieving Immunogenicity | Up to Approximately Week 37
  Immunogenicity is defined the percentage of participants with ADA and neutralizing anti-drug antibodies (nAb).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (8):
  - Lucile Packard Children's Hospital /ID# 240854, Palo Alto, California
  - Nicklaus Children's Hospital /ID# 241174, Miami, Florida
  - New York Medical College /ID# 239208, Valhalla, New York
  - Levine Children's Hospital /ID# 242765, Charlotte, North Carolina
  - Cincinnati Childrens Hospital Medical Center /ID# 239823, Cincinnati, Ohio
  - Children's Hospital of Philadelphia - Main /ID# 239294, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital /ID# 239184, Memphis, Tennessee
  - University of Texas Southwestern Medical Center /ID# 240892, Dallas, Texas
- Australia (3):
  - Children's Hospital at Westmead /ID# 240091, Westmead, New South Wales
  - Royal Children's Hospital /ID# 240384, Parkville, Victoria
  - Perth Children'S Hospital /ID# 240382, Perth, Western Australia
- Universitair Ziekenhuis Leuven /ID# 242384, Leuven, Vlaams-Brabant, Belgium
- Canada (2):
  - Hospital for Sick Children /ID# 240767, Toronto, Ontario
  - CHU Sainte-Justine /ID# 240766, Montreal, Quebec
- Czechia (2):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 239956, Brno, Brno-mesto
  - Duplicate_Fakultni Nemocnice v Motole /ID# 239957, Prague
- France (4):
  - CHU Bordeaux - Hopital Pellegrin /ID# 240832, Bordeaux, Nouvelle-Aquitaine
  - CHU de Nantes, Hotel Dieu -HME /ID# 240831, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy /ID# 240966, Villejuif, Val-de-Marne
  - Hospices Civils de Lyon /ID# 240834, Lyon
- Germany (3):
  - Universitaetsklinikum Erlangen /ID# 240861, Erlangen, Bavaria
  - Universitaetsklinikum Giessen und Marburg /ID# 240787, Marburg, Hesse
  - Universitaetsklinikum Muenster /ID# 239970, Münster, North Rhine-Westphalia
- Israel (3):
  - Schneider Children's Medical Center /ID# 240171, Petah Tikva, Central District
  - Rambam Health Care Campus /ID# 240037, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 240670, Ramat Gan, Tel Aviv
- Italy (3):
  - Azienda Ospedaliero Universitaria Meyer /ID# 240049, Florence, Firenze
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo /ID# 245592, Monza, Monza E Brianza
  - Ospedale Pediatrico Bambino Gesù /ID# 240039, Rome, Roma
- Japan (5):
  - NHO Nagoya Medical Center /ID# 246680, Nagoya, Aichi-ken
  - Kyoto University Hospital /ID# 246907, Kyoto, Kyoto
  - Osaka City General Hospital /ID# 246906, Osaka, Osaka
  - National Cancer Center Hospital /ID# 246722, Chuo-ku, Tokyo
  - National Center for Child Health and Development /ID# 246658, Setagaya-ku, Tokyo
- South Korea (2):
  - Seoul National University Hospital /ID# 239894, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 239895, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Sant Joan de Deu /ID# 240719, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 240715, Barcelona
  - Hospital Infantil Universitario Nino Jesus /ID# 240717, Madrid
- National Taiwan University Hospital /ID# 242890, Taipei City, Taipei, Taiwan
- Koc Universitesi Hastanesi Translasyonel Tıp Arastırma Merkezi /ID# 240026, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No